CLINICAL TRIAL: NCT05516654
Title: Type VI Secretion System in Klebsiella Pneumoniae Relation to Antibiotic Resistance and Biofilm Formation
Brief Title: Type VI Secretion System in Klebsiella Pneumoniae
Acronym: Klebsiella
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Noha Saber Shafik, lecturer of Medical Microbiology and Immunology, faculty of medicine, Sohag University
Other Study IDs: Soh-Med-22-8-23
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Detection of Type VI Secretion System in K.Pneumoniae; Detection of Relation to Ab Resistance, Biofilm
Keywords: Type IV; secretion system; Klebsiella Pneumoniae

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Samples(pus, urine, blood, peritoneal fluid) will be collected from different departments at Sohag university hospital
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Routine bacteriological cultures — culture of different samples on different culture media as nutrient agar, blood agar, MacConkey agar, EMB agar, TSI
Diagnostic Test: Identification of the organism and antibiotic sensitivity will be done by VITEK II — Automated identification of the organism and antibiotic sensitivity will be done by VITEK II
Diagnostic Test: Detection of biofilm formation — Detection of Biofilm formation to the collected organism by tissue culture plate method.
Diagnostic Test: Molecular detection by PCR — Molecular detection of Type VI Secretion System genes, capsular serotyping( k1, k2), and FimH genes by PCR.

SUMMARY:
Klebsiella pneumoniae (K. pneumoniae) is an important opportunistic pathogen contributing to nosocomial and antimicrobial-resistant infections. The increasing prevalence of infections caused by multidrug-resistant K. pneumoniae has emerged as a major clinical and public health threat, while the serous organ and life-threatening infections caused by highly virulent K. pneumoniae have also emerged( Russo and Marr, 2019; Wyres et al., 2020).

DETAILED DESCRIPTION:
Both drug-resistant and highly virulent K. pneumoniae have brought major challenges to clinical treatment and stimulated interest in studying K. pneumoniae. However, knowledge of the genomics, ecology, and pathogenicity of K. pneumoniae is relatively limited. Recently, the type VI secretion system (T6SS) was identified as a virulence factor in K. pneumoniae (Martin and Bachman, 2018). Furthermore, K. pneumoniae was found to exploit the T6SS nano-weapon to destroy bacterial competitors and fungi (Storey et al., 2020).

The bacterial Type VI Secretion System (T6SS) is a membrane-attached contractile phage tail that is physically and Mechanistically similar to a membrane-linked intracellular contractile phage tail. T6SS spike and tube elements, as well as anti-bacterial and anti-eukaryotic effectors, are propelled out of predatory T6SS positive cells and into target cells by a fast conformational shift in the structural framework of a sheath protein complex, according to recent research (Kudryashev et al., 2015).

However, the limited studies and lack of information on the T6SS in K. pneumoniae necessitate further exploration to clarify the physiological metabolism and pathogenic information of this clinically important bacterial species.

ELIGIBILITY:
Inclusion Criteria:

* All patients suffering from infections that can be caused by Klebsiella Pneumoniae.

Exclusion Criteria:

* Samples diagnosed to have organisms other than Klebsiella Pneumoniae

Ages: 12 Weeks to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: -Samples(pus, urine, blood, peritoneal fluid) will be collected from different departments at Sohag university hospital.
  Clinical Data will be obtained as:
  1. Data about clinical manifestations including fever, expectoration, pus from wounds, and diarrhea, urinary symptoms, symptoms of upper respiratory tract infections, symptoms of spontaneous bacterial peritonitis.
  2. Laboratory investigation:
     A-CBC B - CRP C- urine analysis D- serum creatinine E - Serum bilirubin F- ALT G -AST
  3. Routine bacteriological cultures will be done.
  4. Automated identification of the organism and antibiotic sensitivity will be done by VITEK II.
  5. Biofilm formation to the collected organism by tissue culture plate method.
  6. Molecular detection of Type VI Secretion System genes ,capsular serotyping( k1, k2) and FimH genes by PCR.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-09-10 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Isolation and identification of Klebsiella Pneumoniae isolated from different samples and determination of their antibiotics profile | 1 september 2022 to 1 November 2022
Detection of Type VI Secretion System In Klebsiella Pneumoniae and its relation to Antibiotic Resistance and biofilm formation | 2 November 2022 to February 2023

CONTACTS AND LOCATIONS:
Overall Officials: Noha S Shfik, lecturer, Principal Investigator — Faculty of medicine, Sohag university
Locations (1):
- Faculty Of Medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No